CLINICAL TRIAL: NCT05542628
Title: Baseline Reference Values for Concussion Assessments in Football
Status: Enrolling by invitation | Type: Observational
Sponsor: Federation Internationale de Football Association (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention included — No intervention included

SUMMARY:
The primary objective is to provide normal concussion assessment references values for use in football.

All National Football Associations participating in The International Football Association Board's additional permanent substitutions trial are requested to provide baseline assessment data from players within their competitions

DETAILED DESCRIPTION:
Concussions represent a subset of traumatic brain injury (TBI), pragmatically described as a "traumatically induced transient disturbance of brain function caused by a complex physiological process". A sports-related concussion (SRC) can result in substantially different outcomes, ranging from no detectable deficits to transient functional impairments or even life-threatening complications. While the immediate effects of most concussions are short-lived, typically resolving within days, athletes who continue to play following a concussive event may increase their risk of developing short-term, medium-term, and long-term consequences.

Diagnosing and determining the severity of a SRC immediately on- or off-field is challenging, especially because clinical signs can evolve after the mechanism of injury. Since combined injuries of the central and peripheral nervous systems are frequent, determining the locus of injury and therefore underlying explanation for symptoms is difficult and often not possible on- or off-field requiring a more focussed examination. Thus, the diagnosis and estimation of injury severity on- or off-field is a major challenge for the personnel performing an assessment. Nevertheless, an immediate, targeted assessment to support clinical decision-making is of great importance and helps to guide the management approach.

Current advice, when a player sustains a confirmed or suspected concussive injury, is to remove them from play immediately and not return to competition or unrestricted training until signs and symptoms have been managed as per relevant guidelines. Follow-up assessment of concussion incidents is recommended to include the Sport Concussion Assessment Tool 5th Edition (SCAT5). The SCAT5 is a standardized tool for use by healthcare professionals in the evaluation of individuals aged 13 years or older, who are suspected of having sustained an SRC. It comprises a neuropsychological test battery that assesses attention and memory function through 8 different domains. For further assessment of neurocognitive deficits and to inform return to play decisions, the Immediate Post-Concussion Assessment and Cognitive Testing tool version 4 (ImPACT) can also provide valuable information. The ImPACT is a computer-based neurocognitive test battery that provides an objective measure of neurocognitive functioning as an assessment aid in the management of concussed individuals aged 12-80 years.

Post-injury assessments can be compared to the player's assessment results from a non-concussed state (baseline assessment), adding more useful information to their interpretation. Unfortunately, many players do not have baseline assessments performed. Therefore, reference values from similar population groups can act as comparator to determine severity and progression of signs and/or symptoms. Reference values are reported in several sports, but values specific to football players are lacking.

The primary objective is to provide normal concussion assessment references values for use in football.

Our hypothesis is that there will be a variation of minor symptoms in non-concussed players.

Secondary objectives are to provide cumulative frequency distribution of the number of symptoms endorsed at baseline, as well as individual symptom endorsement. Additionally, we aim to provide an overview of cut-off scores and classification ranges to create a reference guide for clinicians of broadly normal and uncommon assessments. Where possible serial baseline assessments will be compared to confirm reliability.

The IFAB additional permanent substitutions trial is expected to run from January 2021 to August 2023 with potential for extension. All teams from participating competitions will be contacted and invited to participate if they have (or expect to) performed baseline assessments within the trial period. Contact information is gathered from the respective competition organisers.

The study is cross-sectional. There are no added procedures which participants have to undertake as being part of the study. The neurocognitive baseline assessments performed should already be a standard component of club practice, in line with international consensus guidelines. Normal practice is that baseline assessments are performed during the pre-season preparation period, at the time of contract commencement for a player entering a new club or one month after having been asymptomatic and medically cleared from a previous concussion injury. Other baseline demographic data will include playing position, age, sex and concussion history. The study will run for the same period as the trial. Early analysis of baseline data can be performed when all competitions have indicated their ability and willingness to participate in this study.

There is a risk of selection bias with potential higher representation of participants competitions with greater resources. To account for this, the study will accept data in any format to reduce the minor burden of participation.

Statistical analysis plan

Demographic data and baseline SCAT5 and ImPACT assessment results are summarized using descriptive statistics according to distribution to provide normal references values. Normal values will be calculated for men and women separately, and according to age, and number of previous concussions. Potential post hoc comparisons between sub-groups will be analysed using independent t-tests or Mann-Whitney U-test according to distributions, and the level of statistical significance will be set at p-value of <0.05.

Sample-size calculation is not performed due to the exploratory study design. We aim to include all available data, but a target of participant data from 1000-2000 players is expected and considered to provide a relevant impression of normal reference values. Data will be analyzed separately for specific federations given sufficient representativeness.

ELIGIBILITY:
Inclusion Criteria:

* Male and female football players from teams in a competition participating in the concussion substitution trial.
* Players without a current suspected or confirmed concussion

Exclusion Criteria:

* Players less than 18 years of age.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The International Football Association Board (IFAB) have initiated a trial of implementing additional permanent concussion substitutions (APCS) for actual or suspected concussions.
  All 211 FIFA member associations (National Football Associations) are invited to participate in this trial. Participation is voluntary. The National football associations can participate with as many competitions as they wish. Competitions refer to different levels of organized leagues, as well as cup tournaments. Additionally, competitions organized by FIFA, such as the FIFA World Cup, are automatically participating in the trial.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
the Sport Concussion Assessment Tool 5th Edition (SCAT5) | through study completion, an average of 2 years.
  The SCAT5 is a standardized tool for use by healthcare professionals in the evaluation of individuals 13 years old or older, who are suspected of having sustained a sports-related concussion. It comprises a neuropsychological test battery that assesses attention and memory function through 8 different domains 1) Symptom number, 2) Symptom severity, 3) Orientation, 4) Immediate memory, 5) Concentration, 6) Neurological examination, 7) Balance errors, 8) Delayed recall.

SECONDARY OUTCOMES:
The Immediate Post-Concussion Assessment and Cognitive Testing tool version 4 (ImPACT) | through study completion, an average of 2 years.
  The ImPACT is a computer-based neurocognitive test battery that provides an objective measure of neurocognitive functioning as an assessment aid in the management of concussion in individuals ages 12-80 years.

CONTACTS AND LOCATIONS:
Locations (2):
- Fèdèration Internationale de Football Association, Zurich, Switzerland
- The University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No